CLINICAL TRIAL: NCT04219865
Title: Study on the Safety, Tolerance and Pharmacokinetics of Single-dose, Increasing and Loading Dose and Maintenance Dose Sequential Intravenous Infusion of Compound Edaravone Injection in Chinese Healthy Volunteers
Brief Title: Safety, Tolerance and Pharmacokinetics Study of Compound Edaravone Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: NJYK-CPEDRV-I
Record Dates: First submitted 2019-12-18; First posted 2020-01-07 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetics
Keywords: Edaravone; Compound edaravone injection

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound Edaravone (Active Comparator): 10 mL per vial (containing edaravone 10 mg and 2-aminoethanesulfonic acid 200 mg)
  Interventions: Drug: Group 1: Compound Edaravone/Placebo Injection; Drug: Group 2: Compound Edaravone/Placebo Injection; Drug: Group 3: Compound Edaravone/Placebo Injection; Drug: Group 4: Compound Edaravone/Placebo Injection; Drug: Group 5: Compound Edaravone/Placebo Injection
- Placebo (Placebo Comparator): 10 mL per vial
  Interventions: Drug: Group 1: Compound Edaravone/Placebo Injection; Drug: Group 2: Compound Edaravone/Placebo Injection; Drug: Group 3: Compound Edaravone/Placebo Injection; Drug: Group 4: Compound Edaravone/Placebo Injection; Drug: Group 5: Compound Edaravone/Placebo Injection

INTERVENTIONS:
Drug: Group 1: Compound Edaravone/Placebo Injection — Compound Edaravone 30mg-600mg (containing edaravone 30 mg and 2-aminoethanesulfonic acid 600 mg) / placebo single intravenous infusion for 30min
Drug: Group 2: Compound Edaravone/Placebo Injection — Compound Edaravone 60mg-1200mg (containing edaravone 60 mg and 2-aminoethanesulfonic acid 1200 mg) / placebo single intravenous infusion for 30min
Drug: Group 3: Compound Edaravone/Placebo Injection — Compound Edaravone 90mg-1800mg (containing edaravone 90 mg and 2-aminoethanesulfonic acid 1800 mg) / placebo single intravenous infusion for 30min
Drug: Group 4: Compound Edaravone/Placebo Injection — Compound Edaravone 120mg-2400mg (containing edaravone 120 mg and 2-aminoethanesulfonic acid 2400 mg) / placebo single intravenous infusion for 30min
Drug: Group 5: Compound Edaravone/Placebo Injection — Maximum tolerated dose of drug / placebo for a single intravenous infusion for 30 minutes three times a day at an interval of 8 h until the last dose on the morning of Day 3, after which the sequential test drug 30 mg-600 mg / placebo will be administered daily from Day 3 night Intravenous infusion, 30 minutes at 12-hour intervals until morning on Day 7

SUMMARY:
Study on the Safety, Tolerance and Pharmacokinetics of Single-dose, Increasing and Loading Dose and Maintenance Dose Sequential Intravenous Infusion of Compound Edaravone Injection in Chinese Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old (including upper and lower limits);
2. Weight ≥50 kg, body mass index (BMI) between 18-28 kg / m2 (including upper and lower limits);
3. Understand and sign the informed consent voluntarily, and volunteer to participate in this research.

Exclusion Criteria:

1. A history of diseases of the heart, liver, lung, kidney, digestive tract, blood, or neuropsychiatric system judged by the investigator as clinically significant;
2. A comprehensive physical examination, neurological examination, laboratory examination, ECG examination, or cognitive assessment indicates that the subject has an abnormality that the researcher has determined to be clinically significant;
3. Have taken any drug within two weeks before the study administration, and the researcher believes that this situation may affect the evaluation results of this study;
4. There is a history of food or drug allergy or allergies that the researcher judges to be clinically significant;
5. Those with positive results of serological examination (HBsAg, anti-HCV, anti-HIV, TP-Ab);
6. A history of alcohol or drug abuse that the investigator believes may affect the evaluation results of this study within one year before the study administration;
7. Cannot quit smoking or drinking during the study period or the carbon monoxide breath test> 7 ppm during the screening period CO breath test, so if the subject's CO breath is> 7ppm, but the urine cotinine test is negative, it means that the CO breath test result may be false positive, the subject can be enrolled;
8. As a subject who has participated in any drug clinical trial within 3 months before the first administration of the study;
9. Those who donated blood or blood products ≥400 mL or 2 units within three months of the study;
10. Do not agree to avoid the use of tobacco, alcohol or caffeinated beverages, or vigorous exercise, or other factors that affect drug absorption, distribution, metabolism, excretion, etc. during the 24 hours before and during the test;
11. Pregnant or lactating women, or those who tested positive for serum HCG before the test administration, or those who were unable or unwilling to take researcher-approved contraception during the study according to the researcher's instructions;
12. Subjects with poor compliance or unable to comply with the relevant provisions of the research protocol due to personal reasons, the investigator judges that the subjects are not suitable to participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) of edaravone and 2-aminoethanesulfonic Acid in single dose groups of compound edaravone injection | 24 hours
Area under curve (AUC) of edaravone and 2-aminoethanesulfonic Acid in multiple doses group after multiple intravenous infusion of compound edaravone injection | 7 Days
Cmax of edaravone and 2-aminoethanesulfonic Acid in single dose groups of compound edaravone injection | 24 hours
Cmax of edaravone and 2-aminoethanesulfonic Acid in multiple doses group after multiple intravenous infusion of compound edaravone injection | 7 Days

SECONDARY OUTCOMES:
Incidence of adverse events of compound edaravone injection | 7 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China